CLINICAL TRIAL: NCT01249287
Title: FMRI in Monitoring Intracerebral Stem Cell Implantation for Chronic Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University Hospital
Other Study IDs: DMR98-IRB-031
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Stroke
Keywords: stroke; stem cell
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A growing number of studies highlight the potential of stem cell transplantation as a novel therapeutic approach for stroke in animal model. But the stem cell therapy for chronic stroke patients has not been well investigated yet. In this study, the investigators will test the hypothesis that intracerebral peripheral blood hematopoietic stem cell (CD34+) (PBSC) transplantation induces neuroplasticity in chronic stroke patients. The remyelination of corticospinal tract in the lesion side, focal increased perfusion and increased cortical activity in the peri-infarcted area will be monitored by the functional MRI after stem cell therapy. The investigators study is aimed to find the potential mechanisms of the functional recovery after stem cell implantation. The investigators also hope to find image surrogate markers for prediction of patient outcome. The possible surrogate markers will be helpful in improving the treatment procedure and patient selection.

ELIGIBILITY:
Inclusion Criteria:

* Old stroke half an year ~3 year
* One-sided MCA infarction
* NIHSS stroke scale: 9-20

Exclusion Criteria:

* Pacemaker
* Cerebral aneurysm clips
* Neurostimulator
* Metallic heart valves
* IUD
* Joint replacement
* Metal plates
* Bone or joint pins
* Vena cava filters
* Embolization coils
* Cochlear implants
* Greenfieid filer
* Seizures
* Claustrophobia
* Bullet/gunshot
* Prosthesis (non-removeable)
* Artificial limbs (non-removeable)
* Surgical slips
* Metal screws or pins>
* Shrapnel/metallic fragments
* Harrington rod
* Insulin pump
* Ever had metal removed from in or around the eye
* Ever been metal worker (i.e., welder, machinist)
* Non-removeable hearing aids
* Birdnest or Gianturco filter
* Pregnant

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-04